CLINICAL TRIAL: NCT03512119
Title: Observational Study of Glucose Tolerance Abnormalities in Patient With Cystic Fibrosis Homozygous for Phe 508 Del CFTR Treated by Lumacaftor-Ivacaftor
Acronym: GLUCORRECTOR
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6403
Record Dates: First submitted 2018-01-15; First posted 2018-04-30 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Cystic Fibrosis Homozygous for Phe 508 Del CFTR; Glucose Intolerance or Newly Diagnosis Diabetes
Keywords: Cystic fibrosis; Glucose tolerance abnormalities; CFTR corrector and potentiator
MeSH Terms: conditions — Glucose Intolerance; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Patient with cystic fibrosis homozygous for Phe 508 del CFTR having a glucose intolerance or newly diagnosis diabetes
  Interventions: Drug: Lumacaftor-Ivacaftor treatment

INTERVENTIONS:
Drug: Lumacaftor-Ivacaftor treatment — Lumacaftor-Ivacaftor treatment during one year

SUMMARY:
Cystic Fibrosis related diabetes (CFRD), a major factor of morbid-mortality in CF, is characterized by a preclinical phase of glucose intolerance particularly long reaching up to 10 years.

At the physiopathology level, insulin secretion is determinant in the glucose tolerance abnormalities in CF. Indeed insulin secretion is dependent of the CFTR activity at the beta cell surface and inhibition of CFTR leads to a decrease in insulin secretion.

Recently, the combination of the lumacaftor, a CFTR corrector, with Ivacaftor, a CFTR potentiator, was studied in patient with CF homozygous for the Phe508 del CFTR mutation patients and showed an improvement of the respiratory state in comparison with the placebo group.

These data suggests that lumacaftor in combination with ivacaftor in targeting CFTR action may have an early impact on the insulin-secretion and consequently on the glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* patients with CF homozygous for the Phe508del CFTR mutation aged 12 years and over
* Combined Lumacaftor-Ivacaftor treatment scheduled or already started
* glucose intolerance in OGTT (ADA criteria) or newly diabetes diagnosed at the OGTT (ADA criteria) or diabetic patients with insulin requirement ≤ 0.3 unit / kg / day or without insulin treatment
* signed informed consent of patient and of one parent OR legal representative for minor subject

Exclusion Criteria:

* hypersensitivity to the active substances or to any of the excipients of Lumactfor -Ivacaftor
* lung and/or liver transplant patient
* Known diabetes with insulin treatment > 0.3 unit / kg / day
* patient pregnant or wishing to pregnancy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with cystic fibrosis homozygous for Phe 508 del CFTR having a glucose intolerance or newly diagnosis diabetes
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Measure of 2 hours plasma glucose value (mmol/l) of OGTT, change from baseline at one year of Lumacaftor-Ivacaftor treatment | Day 0 (traitement beginning) and year 1

SECONDARY OUTCOMES:
Fasting and one hour glucose value of OGTT (mmol/l) | Day 0 (traitement beginning) and year 1
C peptide and insulin values at T0, 1 , 2 hours of OGTT (µg/l) | Day 0 (traitement beginning) and year 1
Glucose, insulin and C peptide AUC of OGTT (µU/L) | Day 0 (traitement beginning) and year 1
HOMA -R , HOMA-S | Day 0 (traitement beginning) and year 1
Mean glucose value per day and 2 h after meal (mg/dl) | Day 0 (traitement beginning) and year 1
Duration in hypoglycemic area [hypo CGM = 2 consecutive values below 3.3 mmol/l - % of time spent] | Day 0 (traitement beginning) and year 1
Duration in hyperglycemic area [for glucose value higher than 7.7 mmol/l, % time /24h] | Day 0 (traitement beginning) and year 1
  Number hypoglycaemic events (below 3.3mmol/L, from midnight to 6 am) Variability glycemic indexes: MAGE (mg/dl), SD (mg/dl)
Number hypoglycaemic events (below 3.3mmol/L, from midnight to 6 am) | Day 0 (traitement beginning) and year 1
  Variability glycemic indexes: MAGE (mg/dl), SD (mg/dl)
Variability glycemic indexes: MAGE (mg/dl), SD (mg/dl) | Day 0 (traitement beginning) and year 1
HbA1c (mmol/l and %) | Day 0 (traitement beginning) and year 1
Daily insulin doses (UI/day) | Day 0 (traitement beginning) and year 1
(BMI) body mass index | Day 0 (traitement beginning) and year 1
Weight (Kg) maximum weight never reached | Day 0 (traitement beginning) and year 1
Albumin and Pre albumin (g/l) | Day 0 (traitement beginning) and year 1
FEV1, Vital Capacity (VC) (L and %) | Day 0 (traitement beginning) and year 1
O2 saturation (%) | Day 0 (traitement beginning) and year 1
Number of cures of antibiotics IV and per os /year and interval between 2 cures (week) | Day 0 (traitement beginning) and year 1

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - Hôpitaux Universitaires de Strasbourg, Strasbourg, Alsace
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Hôpital Renée Sabran, Giens
  - Centre Hospitalier Lyon Sud, Lyon
  - Hôpital NORD - Assistance Publique Hôpitaux de Marseille, Marseille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Hôpital Robert Debré, Paris
  - American Memorial Hospital, Reims
  - Clinique "Mucoviscidose" Presqu'île de Perharidy, Roscoff
  - Hôpital Charles Nicolle, Rouen
  - Hôpital FOCH, Suresnes
  - Hôpital Bretonneau - CHRU de Tours, Tours
  - Hôpital de Clocheville - CHRU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No